CLINICAL TRIAL: NCT05403567
Title: Video Gaming for Home-Based Rehabilitation: Feasibility for Children With Hemiplegic Cerebral Palsy Living in Costa Rica
Brief Title: Video Gaming for Home Rehabilitation for Children With Hemiplegic Cerebral Palsy in Costa Rica
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Universidad de Costa Rica (Other)
Responsible Party: Principal Investigator, Elaine Biddiss, Senior Scientist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0318
Record Dates: First submitted 2022-04-01; First posted 2022-06-03 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: home rehabilitation; upper limb; videogame; mixed methods

STUDY DESIGN:
Masking Description: Outcome Assessor for primary outcome measure is blinded to the time of assessment (eg., baseline, pre-intervention, intervention or post-intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bootle Blast Intervention (Experimental): Children will play the Bootle Blast game at home for 8 continuous weeks.
  Interventions: Other: Bootle Blast Home Intervention

INTERVENTIONS:
Other: Bootle Blast Home Intervention — Children will play BB at home for 8 continuous weeks. Participants will be asked to stop playing at the end of week 8 and the game will be programmatically locked to prevent further play until the post-intervention interviews and assessments are complete.
  Other Names: Bootle Blast Program

SUMMARY:
Economic and geographic barriers can limit access to rehabilitation therapies for children with cerebral palsy (CP). These barriers are magnified in developing countries like Costa Rica, where 43% of children with disabilities do not have access to basic health services. To address this accessibility gap, effective and engaging approaches are needed to motivate and support children in practicing motor therapies at home.

Bootle Blast (BB) is a low-cost, movement-tracking video game that encourages upper limb (UL) exercises at home. BB is mixed-reality; using real-life objects (e.g., toys) in gameplay to target fine motor skills. It is customizable to diverse abilities and therapy goals. BB applies best practices in video game design, theories of motivation and motor learning, to optimize engagement and clinical effectiveness.

This mixed-methods study will assess the feasibility of a family-centred BB home intervention among children with hemiplegic CP. The investigators will address four areas of feasibility to 1) Understand the demand for the BB intervention (i.e., expressed interest in the program), 2) Establish probable efficacy for clinical outcomes related to UL function, activity, and participation, 3) Evaluate implementation of the 8-week BB intervention and 4) Explore acceptability (e.g., participants' experiences).

Fifteen children with a diagnosis of hemiplegic CP (7-17 yrs) and one of their primary caregivers will participate. This study consists of three phases, each one contributing to the development of the next one. In Phase 1 (demand), recruitment rates and percentage of children with appropriate in-home technology to play will be collected during screening. A pre-intervention interview will explore participants' expectations for the intervention. In Phase 2, study assessments will be performed via videoconference (probable efficacy). Measures will target UL activity and related participation. Children will play BB at home for 8 weeks. Computer-system logs and data from reported technical barriers will be collected (implementation). In Phase 3 parents and children will participate in a post-intervention interview to explore their experiences and perceived value of the BB program (acceptability).

Worldwide, children face accessibility barriers to motor therapy services. This study will provide learnings on how therapy gaming interventions can/should be implemented to bridge accessibility gaps, engage children and improve access to care.

DETAILED DESCRIPTION:
RESEARCH QUESTION AND OBJECTIVES This feasibility study will use a multi-stage mixed methods design20. It aims to address the possibility of successfully implementing the BB program intervention in a small scale, semi-controlled, real-world environment among Costa Rican families with children with hemiplegic CP. It will address our overall research question: To what extent is a video game designed for upper limb therapy (BB) feasible for use in a home rehabilitation program for children with hemiplegic CP in Costa Rica who experience barriers accessing therapy services? In this study, the investigators are particularly interested in four areas of feasibility: demand, implementation, limited-efficacy testing and acceptability as defined by Bowen et al17. Demand looks at the extent to which an intervention is likely to be used in a given setting or population. Implementation evaluates the extent to which the intervention can be implemented as proposed. Limited-efficacy aims to inform the potential of the intervention in a limited way (e.g., convenience sample). Acceptability focuses on how participants react to the intervention.

To address our research question, our specific objectives are:

1. To understand demand for the BB intervention, including expressed interest in the program, capacity to integrate BB into the family home and routine, and the expectations of children with hemiplegic CP and their parents for the BB intervention.

   Indicators:
   * Recruitment rate of 3 child-parent dyad a month for 5 months (n=15), with a ≥10% response rate (i.e., expressed interest, fit the eligibility criteria)
   * At least 80% of families who wish to participate will have an appropriate screen and space to play BB.
   * The family-directed play time goal, which is sensitive to family schedules and routines, provides a "therapy dose" that could reasonably be expected to be clinically meaningful [i.e., at least 45 minutes a week13].
   * The family can define at least one therapy goal that aligns with the scope of the BB intervention.
   * Identify the expectations that children and their parents have of the BB program (e.g., improving in a meaningful activity involving the upper limb, having a fun alternative to exercise their hands/arms).
2. To establish limited efficacy by measuring pre-post intervention changes in clinical outcomes related to upper limb function, activities and participation in children with hemiplegic CP using BB for 8 weeks at home.

   Indicators:

   ● At least 75% of the children will show clinically meaningful improvements from pre- to post-intervention16 in: a) one of the dimensions of the Quality of Upper Extremity Skills Test (QUEST)the and/or, b) perceived performance on a self-identified upper limb goal area as measured by the Canadian Occupational Performance Measure (COPM)20. Secondary outcome measures are detailed in the methods section.
3. To evaluate implementation of the 8-week BB home intervention among children with hemiplegic CP, including ability to meet family-directed play time goals.

   Indicators:
   * ≥80% of children will a) achieve their weekly play time goal in at least 6 out of the 8 weeks, and b) complete the 8-week intervention.
   * Number and type of reported technical barriers.
   * ≤20% of participants will experience a technical barrier which will prevent use of the system for more than 4 days (e.g., technical difficulties will be easy to overcome with phone/video assistance).
4. To explore acceptability of the BB intervention through children's and parents' game and therapy related experiences

Indicators:

• To explore the perceived value of the intervention by children and their parents, including factors related to motivation1, the modality of therapy (i.e., home based), the use of the family-centered approach (e.g., family-directed play time goal), and the barriers they face accessing therapy services.

These feasibility success criteria were developed with reference to previous studies of similar upper extremity, home-based interventions in children with CP8,16,18

OVERVIEW OF STUDY DESIGN Two teams of researchers (Universidad de Costa Rica - HB, appendix M - research team) will carry out this study. This study follows an advanced multistage mixed methods design framework, with three sequential stages of data collection21 detailed in three phases. Each phase will address a specific objective.

Phase 1 - Demand [QUAL (quant)] : This phase addresses objective one and involves both a quantitative and a qualitative component. Data on recruitment rates, and access to appropriate space and technology to play indicators (quant) will be collected at the screening stage. Additionally, eligible children and their parent will be interviewed to establish their expectations for the BB intervention, and to understand how/if the intervention can be tailored to the family's needs and context (QUAL). Data collected in this phase will inform sampling and the intervention design for phase two. For example, if a family's expectations for the intervention do not align with what can be achieved by participating in the BB program, then they will not be included in the intervention phase (phase 2). Data from the semi structured interview from eligible participants will also be used to tailor the intervention in a family-centred way, to maximize potential for positive outcomes. For example, defining a realistic play time goal that aligns with the family's schedule and context.

Phase 2 - Limited Efficacy and Intervention [QUANT (qual)]: In this phase, 15 children-parent dyads will be provided with BB to play at home for 8 continuous weeks, and the necessary computer system to use it, namely the Orbbec Persee14. In phase two, children and parents will also participate in a weekly videocall (Zoom) where several research clinical assessments will be evaluated(QUANT Additionally, during the 8-week intervention a monitoring therapist (qual) will perform weekly 15-minute check-in video calls to each participant. During these video calls a short video assessment will also be conducted (Perceived Quality Rating Scale, PQRS). Data collected in Phase 2 related to play adherence, reported technical barriers, and field notes from the monitoring therapist will be used to inform and better guide the conversations during the post-intervention interviews in phase 3. For example, if a marked increase or decrease in play was observed at different time points in the intervention, this might be explored in further detail in the post-intervention interview.

Phase 3 - Acceptability [QUAL]: This strand will adopt a qualitative descriptive approach21 in order to explore participants' experiences about the intervention via a semi-structured, post-intervention interview. Analysis of these data will be used to better understand the results from the clinical research assessments. Additionally, the investigators will identify the extent to which family expectations for the BB intervention (established in the pre-interview phase) aligned with the experiences reported in the post-interviews during phase 3.

In rehabilitation clinical practice it is impractical to separate clinical outcomes from the social environment of the patient. The nature of this work calls for a mixed methods research approach since the quantitative and qualitative components cannot stand alone, and need to be integrated to fully answer the research question22. Data from each phase will be first analyzed separately and then brought together for analysis and comparison. Appendix F visually details how the data generated in each phase will be integrated to address our specific research objectives.

MIXED METHODS ANALYSIS AND INTEGRATION Integration will occur at the design, methods, interpretation and reporting levels. Members of the research team involved in the integration of results include researchers with clinical background in childhood disability, quantitative and/or qualitative expertise. At the methods level, the study uses a mix of connecting, building and merging approaches20. Integration using a contiguous approach will be used at the interpretation and reporting levels20. Appendix F visually details how each objective informs/links to each other at different integration levels.

Phase 1 and 2: A sample of participants from phase 1 will be selected to participate in phase 2, following the process and criteria described in the participants sections. Second, preliminary analysis from the pre-intervention interviews (phase 1) will be used to individually tailor the BB intervention in a family-centred way to maximize potential for positive outcomes in phase 2.

Phase 2 and 3: Field notes from the weekly phone calls and results from the computes logs from phase 2 will be used to better guide the conversation during the semi-structured interview with each participant in phase 3. For example, if a marked increase or decrease in play was observed at different time points during the intervention, if a participant reported technical barriers and/or an increase in play motivation during some of the weeks, this can be explored in further detail in the post-intervention interview.

Additionally, results from both phases will be brought together for interpretation. Quantitative and qualitative results will be merged to better understand changes in hand/arm clinical outcomes, contextual factors that influenced the results of the intervention, detailed information about the nature of the experience of the participants, and development of recommendations that might be necessary for future real-world implementation of similar interventions.

Phase 1 and 3: Results from both phases will be brought together to identify the extent to which the family expectations for the intervention in phase 1 coincide and/or align with the experiences reported in phase 3.

Integration with a contiguous approach will be used for all phases at the interpretation and reporting levels, where results from each phase will first be presented separately, and then interpret together in the discussion section to answer our research question20. Intention to maintain rigour in this mixed methods proposal has been addressed by following the GRAMMS guidelines48.

IMPACT Worldwide, children face accessibility barriers to motor therapy services. This study will provide valuable learnings on how low-cost therapy gaming interventions (like BB) technologies, such as motion-based video games, can/should be implemented to bridge accessibility gaps and improve access to rehabilitation for children with PC. The focus on the patient and family-centered approach of this project also intends to facilitate knowledge translation and dissemination of results to the community with PC, since for these families the results of research studies can generally be difficult to generalize.

Video games such as BB can facilitate access to therapy for children with PC, especially for those living in low-income families and / or rural areas. This aligns with the international right of children to access adequate medical care, and with Costa Rica's public policy regarding disability and child health care. Study results will also inform future work to establish BB as an effective, accessible, and fun option for upper-limb home rehabilitation in developing countries. For our particular project and as per the Costa Rican bioethical law, children who complete the 8 week-intervention will keep the BB video game and the necessary computer system to play it.

ELIGIBILITY:
Participants: Children and parent dyads living anywhere in the country can participate in this phase. Dyads will be screened to participate in the pre-intervention interview according to the following criteria:

Inclusion Criteria:

* Diagnosis of hemiplegic CP.
* 7 to 17 years of age: This age range was selected given the popularity of video games for children at this stage. This age group in CP has been studied successfully in previous research focused on active video game play, showing potential for change across their motor outcomes8-10.
* Motor impairment of the upper limb: difficulty to manipulate objects and/or perform activities of daily living with one hand/arm in alignment with the Manual Classification System levels I-III18, as reported by the parent and assessed via telephone by the clinician-researcher (DC - Appendix B, telephone screening). These children would require minimal assistance in playing the video game in the home environment.
* Having a primary family caregiver willing to participate.
* Resident of Costa Rica.
* Child and parent are able to understand and communicate verbally in Spanish or English.
* Child and/or parent are able to read and write.
* Child and/or parent has knowledge on how to use email and receive a video call or have a support person willing to assist them during the clinical assessment processes.
* Child and/or parent has access to a cellphone or computer at home.
* Ability to cooperate, understand, and follow simple instructions for game play as reported by parent.
* Having a TV screen (or similar) at home.
* Having an accessibility barrier that currently limits their access to upper limb rehabilitation services. These barriers include but are not limited to: the family is unable to pay for therapy, services are not available in their living area, or there is a lack of adapted transportation for the child to travel to a therapy center, as reported by the caregiver.

Exclusion Criteria:

* Receiving hand and arm therapy at the time of intervention.
* History of uncontrolled epilepsy. If the child has a history of epilepsy, they will require a note from a doctor indicating it would be safe to play video games as required in this study. A note will not be required if the child currently engages in at least 30 minutes of screen time a day on 2 or more days in a week as documented by a primary caregiver.
* Visual or hearing impairments that limit the ability to play the video game.
* Has received constraint induced movement therapy in the past 6 months, or botulinum toxin injections, or active therapy of the upper extremity within three months of the study enrollment.
* History of upper limb injury or disability that would make light exercise unsafe as reported by the caregiver.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Upper Extremity Skills Test (QUEST) | weeks 4 & 5 (pre assessment sessions), week 15 (post assessment session)
  The QUEST is a 34-item criterion-referenced observation test with four domains: dissociated movement, grasp, weight-bearing, and protective extension. Domain scores are a summed item score which is converted into a standardized percentage. The total score is an average of the domain scores with higher scores indicating increased levels of achievement. The reliability and the concurrent validity for the study population is well established. For the purposes of this research study, only the dissociated movement and grasp domains will be used as the weight-bearing and protective extension dimensions may be more difficult to capture over Zoom. The minimally clinically important difference (MCID) for the QUEST is reported as a positive change of 4.89 score units on any dimension. The QUEST requires a chair and table to sit at, four 1" cubes, a cup, a pencil or crayon, blank paper and cheerios.
Change in Canadian Occupational Performance Measure (COPM) | week 5 (pre assessment session), week 15 (post assessment session)
  The COPM evaluates the performance, and the satisfaction with performance of self-identified therapy goals. Participants will first identify hand/arm goals of daily life activities that they wish to improve (e.g., cutting with fork and knife). Parent and child will rate together the child's level of performance and satisfaction with performance over a 10-point numerical scale (1 is poor/low and 10 is high/good) for each of their identified goals. This measure has shown good reliability, construct validity and responsiveness for use with children with CP. A change of 2 points is considered a minimal clinically important response

SECONDARY OUTCOMES:
Active Range of Motion (aROM) | weeks 4 & 5 (pre assessment sessions), week 15 (post assessment session)
  Is a foundational measure for associated changes in function. Manual goniometry has good test-retest reliability (ICC>0.8) and moderate-to-good inter-rater reliability for the wrist and elbow in children with CP. A minimal detectable difference of 5 degrees has been reported in children with spastic CP. In recent years, the potential of goniometer applications that rely on 2D video analysis has been established. A virtual goniometer from an open-source, 2D motion analysis software (Kinovea) will be used to measure aROM of the shoulder, elbow and wrist joints of the child's affected upper limb. aROM data will be measured from the QUEST dissociated movement videos.
Change on the Performance Quality Rating Scale (PQRS) | weekly throughout study completion, on average 15 weeks
  The PQRS is an observational, video-based tool that looks at actual performance on client-selected activities. It has been used with children with diverse diagnoses, including CP. It uses a 10-point scale with a score of 1 indicating ''can't do the skill at all'' and 10 indicating ''does the skill very well". Judgement of quality includes timeliness of completion, accuracy, safety, and overall quality of performance or product. Ratings are based on an average of completeness and quality. Inter-rater reliability is moderate (0.71-0.77). Test-retest reliability is excellent (>0.9) across time periods and multiple raters. The average smallest detectable difference is 2.55. The MCID has not yet been established for the PQRS. Internal responsiveness is high with large effect sizes reported. Of note, the PQRS and COPM can complement each other, based on their objective / subjective nature, and therapeutic evaluation versus participant's perception.
Change on the Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) | weeks 4 & 5 (pre assessment sessions), week 15 (post assessment session)
  Includes the assessment of: active and passive range of motion, tone, performance of activities of daily living (client reported) and evaluation of 16 activities using the hand and arm. The SHUE focus on the fingers, hand and elbow movements. All the assessments are video recorded and scored at a later time. For this study, we will only assess the 16 hand and arm tasks, since evaluating tone is not possible via Zoom, range of motion will be assessed using the QUEST, and performance of activities of daily living is captured by the COPM.
  The 16 hand and arm activities are evaluated based on the dynamic segmental alignment (DSA) and the spontaneous functional analysis (SFA) of the involved upper extremity. The scoring uses a modified house scale from 0-5 for the SFA, and 0-3 for the DSA, where 0 is the lowest / less functional score. The SHUEE has excellent validity and reliability for both, the DSA and the SFA components in children with hemiplegic CP.
Change in the Box and Blocks Test (BBT) | weeks 4 & 5 (pre assessment sessions), week 15 (post assessment session)
  The test consists of a wooden box with two compartments with a vertical division and 150 small cubes. Measures unilateral gross manual dexterity by asking the participant to pass the maximum number of cubes possible above the division, from one side to another, in 60 seconds. The test takes 2 to 5 minutes to complete and is appropriate for ages 6 and up. BBT has excellent test-retest reliability, inter- and intra-rater reliability, high responsiveness, and criterion and construct validity in typically developing children and adults of diverse diagnoses. The MCID reported for children with CP is 1.9 (blocks) on the more affected hand and 3.0 (blocks) on the less affected hand. For this project a modified kit will be sent to the participant's home, consisting of a cardboard box instead of a wooden box (original box dimensions will be kept).
Change on the Children's Hand-Use Experience Questionnaire | week 4 (pre assessment session), and week 15 (post assessment session)
  Aims to capture the perceived quality and effectiveness of the child's use of their affected hand in bilateral task performance against 29 activities. The results are transformed by means of Rasch analysis to a 0-100 unit scale placed on rulers. The rulers demonstrate how the hand works (0=does not use the hand at all, 100= uses the hand very well); the time it takes for the child to perform the activity in relation to peers (0= takes a lot more time, 100= takes the same amount of time) and how bothered the child is about the decreased hand function (0=it bothers the child a lot, 100= it does not bother the child). The result in the report is a summary of the ratings. This self-reported measure can be completed by the child or the parent. For the purposes of this study, we will ask the caregiver to complete this measure.
Count of number of intentional therapeutic movements achieved during active and passive playtime. | Weeks 1 to 8 during the intervention
  BB records all user activity within the game (e.g. games played, etc.). Active (e.g. focused on therapeutic movement) and passive (e.g. navigating menus) playtime and the number of intentional therapeutic movements achieved (e.g. arm reach, cross-body reach) will be recorded. Of note, video recordings collected via Bootle Blast are for the most part non-identifying. The face and much of the background, with the exception of that immediately surrounding the player, are blocked out to preserve privacy.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (2):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada
- Universidad de Costa Rica, San Pedro, Provincia de San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilde PE, Kliim-Due M, Rasmussen B, Petersen LZ, Petersen TH, Nielsen JB. Individualized, home-based interactive training of cerebral palsy children delivered through the Internet. BMC Neurol. 2011 Mar 9;11:32. doi: 10.1186/1471-2377-11-32. PMID 21392370
- [Background] Biddiss E, Chan-Viquez D, Cheung ST, King G. Engaging children with cerebral palsy in interactive computer play-based motor therapies: theoretical perspectives. Disabil Rehabil. 2021 Jan;43(1):133-147. doi: 10.1080/09638288.2019.1613681. Epub 2019 May 19. PMID 31104517
- [Background] Fetters MD, Curry LA, Creswell JW. Achieving integration in mixed methods designs-principles and practices. Health Serv Res. 2013 Dec;48(6 Pt 2):2134-56. doi: 10.1111/1475-6773.12117. Epub 2013 Oct 23. PMID 24279835
- [Background] Romeiser-Logan L, Slaughter R, Hickman R. Single-subject research designs in pediatric rehabilitation: a valuable step towards knowledge translation. Dev Med Child Neurol. 2017 Jun;59(6):574-580. doi: 10.1111/dmcn.13405. Epub 2017 Feb 22. PMID 28224606
- [Background] Cusick A, Lannin NA, Lowe K. Adapting the Canadian Occupational Performance Measure for use in a paediatric clinical trial. Disabil Rehabil. 2007 May 30;29(10):761-6. doi: 10.1080/09638280600929201. PMID 17457734
- [Background] Martini R, Rios J, Polatajko H, Wolf T, McEwen S. The performance quality rating scale (PQRS): reliability, convergent validity, and internal responsiveness for two scoring systems. Disabil Rehabil. 2015;37(3):231-8. doi: 10.3109/09638288.2014.913702. Epub 2014 Apr 28. PMID 24766150
- [Background] Skold A, Hermansson LN, Krumlinde-Sundholm L, Eliasson AC. Development and evidence of validity for the Children's Hand-use Experience Questionnaire (CHEQ). Dev Med Child Neurol. 2011 May;53(5):436-42. doi: 10.1111/j.1469-8749.2010.03896.x. Epub 2011 Mar 17. PMID 21413973
- [Derived] Chan-Viquez D, Fernandez-Huertas H, Montserrat-Gonzalez C, Khan A, Fehlings D, Munce S, Wright FV, Biddiss E. Feasibility of a home-based home videogaming intervention with a family-centered approach for children with cerebral palsy: a randomized multiple baseline single-case experimental design. J Neuroeng Rehabil. 2024 Sep 4;21(1):151. doi: 10.1186/s12984-024-01446-2. PMID 39227911